CLINICAL TRIAL: NCT03206138
Title: A Randomized, Open-label Study to Evaluate the Safety and Efficacy of GX-188E, a DNA Therapeutic Vaccine Administered Intramuscularly by Electroporation, With GX-I7 Intravaginal Application or Imiquimod Topical Application in HPV16 and/or 18 Positive Patients With CIN3.
Brief Title: Safety and Efficacy of GX-188E Administered Via EP Plus GX-I7 or Imiquimod.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Collaborators: Genexine, Inc. (Industry)
Responsible Party: Principal Investigator, Jongsup Park, Professor, Seoul St. Mary's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GX-188E_GX-I7_IMQ_CIN3
Record Dates: First submitted 2017-06-20; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Cervical Intraepithelial Neoplasia 3
Keywords: Investigator trial; Cervical Intraepithelial Neoplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — efineptakin alfa; Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GX-188E, GX-I7 (Experimental): GX-188E + GX-I7
  Interventions: Biological: GX-188E, GX-I7
- GX-188E, Imiquimod (Experimental): GX-188E + Imiquimod
  Interventions: Biological: GX-188E, Imiquimod

INTERVENTIONS:
Biological: GX-188E, GX-I7 — Experimental: 1mg of GX-188E administered IM using EP device 3 times and 3mg of GX-I7 administered in cervix 4 times.
  Arms: GX-188E, GX-I7
Biological: GX-188E, Imiquimod — 1mg of GX-188E administered IM using EP device 3 times and 12.5mg of Imiquimod application at cervix 8 times.
  Arms: GX-188E, Imiquimod

SUMMARY:
This is a study to investigate the safety and efficacy of GX-188E administered IM plus local administration of GX-I7 or Imiquimod at cervix in subjects with cervical intraepithelial neoplasia (CIN) 3.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to comply with all study procedures and voluntarily signs informed consent form.
* Female subjects age 19-50 years.
* HPV 16 and/or 18 positive.
* Colposcopy is satisfactory based on visualization of the entire squamocolumnar junction and the upper limit of the entire aceto-white or suspected CIN disease area
* Histopathologically diagnosed with Cervical Intraepithelial Neoplasia 3, CIN 3.

Exclusion Criteria:

* Pregnancy or breastfeeding
* History of previous therapeutic HPV vaccination (individuals who have been immunized with licensed prophylactic HPV vaccines are not excluded).
* Positive serological test for hepatitis C virus or hepatitis B virus surface antigen (HBsAg) or human immunodeficiency virus (HIV).
* Any other ineligible condition at the discretion of the investigator that would be ineligible to participate the study.

Ages: 19 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-05-30 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Ratio of subjects who have histopathological regression of cervical lesions to CIN 1 or less in HPV 16 or 18-associated CIN3 subjects. | at week 20

SECONDARY OUTCOMES:
Ratio of subjects with clearance of HPV 16 or 18 and histopathological regression of cervical lesions to CIN 1 or less. | at week 20, and week 36
The change of cytology of uterine cervix compared to baseline. | at screening, week 12, week 20, and week 36
Flt-3L concentrations in blood samples. | at week 14, week 20, and week 36.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul St. Mary's hospital, Seoul, South Korea